CLINICAL TRIAL: NCT01178281
Title: A Phase-3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Compare Efficacy and Safety of Pomalidomide in Subjects With Myeloproliferative Neoplasm-Associated Myelofibrosis and Red Blood Cell-Transfusion-Dependence
Brief Title: Study of Pomalidomide in Persons With Myeloproliferative-Neoplasm-Associated Myelofibrosis and RBC-Transfusion-Dependence
Acronym: RESUME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-4047-MF-002; 2010-018965-42 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-08-10 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Primary Myelofibrosis; MPN-associated Myelofibrosis
Keywords: Myelofibrosis; Post-polycythemia vera myelofibrosis; Post-essential thrombocythemia myelofibrosis; RBC-transfusion-dependence; Primary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — pomalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pomalidomide 0.5 mg (Experimental): Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects or disease progression.
  Participants who were RBC-transfusion independent or experienced clinical benefit (defined as a reduction from Baseline of ≥ 50% in RBC-transfusion frequency during the prior 84-day interval) could continue to receive pomalidomide until loss of RBC-transfusion independence response or clinical benefit, or other criteria for treatment discontinuation applied.
  Interventions: Drug: Pomalidomide 0.5 mg
- Placebo (Placebo Comparator): Participants received placebo taken by mouth once daily for at least 168 days unless there were unacceptable side effects or disease progression.
  Participants who were RBC-transfusion independent or experienced clinical benefit could continue to receive placebo until loss of RBC- transfusion independence response or clinical benefit, or other criteria for treatment discontinuation applied.
  Interventions: Drug: Placebo
- China Extension: Pomalidomide 0.5 mg (Experimental): Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects, disease progression, or they received a RBC-transfusion.
  Participants who experienced anemia response could continue treatment until the response was lost or other criteria for treatment discontinuation applied.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide 0.5 mg — Pomalidomide 0.5 mg capsule taken by mouth once daily. Immunomodulatory agent with demonstrated efficacy in the treatment of subjects with RBC-transfusion-dependence associated with MNP-associated myelofibrosis.
  Other Names: CC-4047; Pomalyst; Imnovid
  Arms: Pomalidomide 0.5 mg
Drug: Placebo — Placebo Comparator to active drug; Placebo capsule taken by mouth once daily
  Arms: Placebo
Drug: Pomalidomide — Pomalidomide 0.5 mg capsule taken by mouth once daily.
  Other Names: CC-4047; Pomalyst; Imnovid
  Arms: China Extension: Pomalidomide 0.5 mg

SUMMARY:
The objective of this study is to determine whether pomalidomide is safe and effective in reversing red blood cell (RBC)-transfusion-dependence in persons with myeloproliferative neoplasm (MPN)-associated myelofibrosis (global study) and in reversing anemia in Chinese with MPN-associated myelofibrosis and severe anemia not receiving RBC-transfusions (China extension study only)

DETAILED DESCRIPTION:
The multicenter global study was conducted in 15 countries including Australia, Austria, Belgium, Canada, China, France, Germany, Italy, Japan, the Netherlands, Russia, Spain, Sweden, the United Kingdom, and the United States. The global study enrolled participants with myeloproliferative neoplasm (MPN)-associated myelofibrosis and RBC-transfusion-dependence. Participants were randomly assigned to receive pomalidomide or placebo in a blinded fashion.

In most countries participating in the global study, RBC-transfusions are typically given for a hemoglobin level <80-90 g/L. In China, RBC-transfusions are rarely given unless the hemoglobin level is <60 g/L. Consequently, few Chinese with MPN-associated myelofibrosis meet RBC-transfusion-dependence criteria of the global study. A China-specific extension was developed to test the ability of pomalidomide to improve severe anemia (defined as a hemoglobin < 80 g/L for ≥ 84 days in persons not receiving RBC-transfusions).

The China-specific extension study consisted of a single-arm, open-label study in adults with MPN-associated myelofibrosis and severe anemia not receiving RBC transfusions with the objective of describing the frequency of anemia response.

The Global (intent-to-treat [ITT] and safety) population in the main study and the China extension (ITT and safety) population are mutually exclusive.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Myeloproliferative-neoplasm (MPN)-associated myelofibrosis
* RBC-transfusion-dependence (global study):

  * Average RBC-transfusion frequency ≥ 2 units/28 days over at least the 84 days immediately prior to randomization. There must be no interval > 42 days without ≥ 1 RBC-transfusion.
  * Only RBC-transfusions given when the hemoglobin ≤ 90 g/L³ are scored in

determining eligibility.

* RBC-transfusions due to bleeding are not scored in determining eligibility.
* RBC-transfusions due to chemotherapy-induced anemia are not scored in determining eligibility.

  * Severe anemia (China-specific extension):
* ≥ 2 hemoglobin concentrations ≤ 80 g/L for ≥ 84 days immediately before the day of enrollment.
* No RBC-transfusion within 6 months prior to enrollment.

  * Hemoglobin ≤ 130 g/L at randomization (global study); ≤ 80 g/L at enrollment in the China-specific extension.
  * Bone marrow biopsy within 6 months (global study only).
  * Inappropriate to receive blood cell or bone marrow allotransplant, erythropoietin and androgenic steroids
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
  * Agree to follow pregnancy precautions as required by the protocol.
  * Agree to receive counseling related to teratogenic and other risks of pomalidomide.
  * Agree not to donate blood or semen.

Exclusion Criteria:

* Prior blood cell or bone marrow allotransplant.
* Use of drugs to treat MPN-associated myelofibrosis ≤ 30 days before starting study drug.
* Treatment with erythropoietin or androgenic steroids ≤ 84 days before starting study drug.
* Anemia due to reasons other than MPN-associated myelofibrosis.
* Pregnant or lactating females.
* More than 10% blasts by bone marrow examination or more than 10% blasts in blood in consecutive measurements spanning at least 8 weeks
* Prior history of malignancies,other than the disease being studied, unless the subject has been free of the malignancy for ≥ 5 years with the following exceptions:

  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T 1a or T 1b using TNM [tumor, nodes, metastasis] clinical staging system)
* Human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections.
* Prior treatment with pomalidomide.
* Allergic reaction or rash after treatment with thalidomide or lenalidomide
* Any of the following laboratory abnormalities:

  * Neutrophils < 0.5x10^9 /L
  * Platelets < 25 x 10^9 /L
  * Estimated glomerular filtration rate (kidney function) < 30 mL/min/1.73 m²
  * Aspartate aminotransferase (AST) and alanine transaminase (ALT) > 3.0 x upper limit of normal (ULN)
  * Total bilirubin ≥ 4 x ULN;
* Uncontrolled hyperthyroidism or hypothyroidism.
* Deep venous thrombosis (DVT) or pulmonary embolus (PE) < 6 months before starting study drug
* Clinically-important heart disease within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Peter P Gale, MD, Ph.D., Study Director — Celgene Corporation
Locations (87):
- United States (17):
  - Mayo Clinic, Scottsdale, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai School of Medicine Brookdale University Hospital, Brooklyn, New York
  - Weill Medical College of Cornell University, New York, New York
  - Ruttenberg Treatment Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Medicine Taussig Cancer Institute, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Avera Hematology and Transplant, Sioux Falls, South Dakota
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Gosford Hospital, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Frankston Hospital, Frankston, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (3):
  - Medizinische Universitatklinik Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Medizinische Universitat Wien, Vienna
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Grand Hopital de Charleroi, Charleroi
  - Universitaire Ziekenhuis Leuven Gathuisberg, Leuven
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal, Montreal
- China (6):
  - Peking University People's Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jiangsu Province Hospital, Jiangsu
  - Shanghai Ruijin Hospital, Shanghai
  - West China Hospital, Sichuan University, Sichuan
  - Blood Disease Hospital Chinese Academy of Medical Sciences, Tianjin
- France (8):
  - Hopital Albert Michallon, La Tronche
  - Hopital Saint Vincent de Paul, Lille
  - CHU Dupuytren, Limoges
  - Hopital Saint-Louis, Paris
  - CHRU - Hopital du Haut Leveque, Pessac
  - Hopitaux Universitaires de Strasbourg, CHU Haute-Pierre, Strasbourg
  - Hopital Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Universitatsklinikum Aachen, Aachen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - Johannes Wesling Klinikum Minden, Minden
  - Universitatsklinikum Ulm, Ulm
- Italy (8):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - Azienda Ospedaliera San Luigi Gonzaga, Orbassano
  - IRCCS Fondazione Policlinico San Matteo, Universita di Pavia, Centro per lo Studio della Mielofibrosi, Pavia
  - IRCCS Fondazione Policlinico San Matteo, Universita di Pavia, Ematologia, Pavia
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese
- Japan (6):
  - Juntendo University Hospital, Bunkyou-ku
  - Kyushu University Hospital, Fukuoka
  - Tokai University Hospital, Isehara
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Tokyo Medical University Hospital, Shinjuku
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Erasmus Medish Centrum, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny im. F.Chopina, Rzeszów
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 PAM, Szczecin
  - Centralny Szpital Kliniczny MSWiA, Warsaw
- Russia (4):
  - Russian Scientific Haematology Centre, Moscow
  - Federal State Institution Russian Scientific-research Institute of Hematology and Transfusiology of Federal Medical-Biological Agency of Russia, Saint Petersburg
  - State Pavlov Medical University, Saint Petersburg
  - Federal State Institution "Federal Centre of Heart, Blood and Endocrinology of Rosmedtechnologies named after V.A. Almazov", Saint Petersburg
- Spain (4):
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Puerta De Hierro Majadahonda, Majadahonda
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Clinico de Valencia, Valencia
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (7):
  - Belfast City Hospital, Belfast
  - Beatson Oncology Centre, Glasgow
  - John Radcliffe Hospital NHS Trust, Headington
  - St. Thomas Hospital, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Tefferi A, Al-Ali HK, Barosi G, Devos T, Gisslinger H, Jiang Q, Kiladjian JJ, Mesa R, Passamonti F, McMullin MF, Ribrag V, Schiller G, Vannucchi AM, Zhou D, Reiser D, Zhong J, Gale RP. A randomized study of pomalidomide vs placebo in persons with myeloproliferative neoplasm-associated myelofibrosis and RBC-transfusion dependence. Leukemia. 2017 Apr;31(4):896-902. doi: 10.1038/leu.2016.300. Epub 2016 Oct 24. PMID 27773929
- [Derived] Begna KH, Pardanani A, Mesa R, Litzow MR, Hogan WJ, Hanson CA, Tefferi A. Long-term outcome of pomalidomide therapy in myelofibrosis. Am J Hematol. 2012 Jan;87(1):66-8. doi: 10.1002/ajh.22233. Epub 2011 Nov 12. PMID 22081489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the global study were enrolled at 72 clinical centers in 15 countries. In addition, the China-specific extension study enrolled participants with myeloproliferative neoplasm (MPN)-associated myelofibrosis and severe anemia not receiving red blood cell (RBC)-transfusions at 5 sites in China.
Pre-assignment Details: Participants in the global study were randomized 2:1 to receive blinded pomalidomide or placebo. All participants in the China extension received open-label pomalidomide. Randomization was stratified by age (≤ vs >65 years), white blood cells (< or ≥25 × 10⁹/L) and baseline transfusion requirement (≤ vs >4 units RBC/28 days over the prior 84 days).
Groups:
- Placebo: Participants received placebo taken by mouth once daily for at least 168 days unless there were unacceptable side effects or disease progression.
  Participants who were RBC-transfusion independent or experienced clinical benefit could continue to receive placebo until loss of RBC-transfusion independence response or clinical benefit, or other criteria for treatment discontinuation applied.
Period: Overall Study
Arm/Group | Pomalidomide 0.5 mg | Placebo | China Extension: Pomalidomide 0.5 mg
Started | 168 | 84 | 15
Received Study Drug | 167 | 83 | 15
Completed (Completed study, no longer in follow-up) | 168 | 84 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all randomized (global study) or enrolled (China extension study) participants
Groups:
- Pomalidomide 0.5 mg: Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects or disease progression. Participants who experienced clinical benefit (defined as a reduction from Baseline of ≥ 50% in RBC-transfusion frequency during the prior 84-day interval) could continue to receive pomalidomide until the definition of clinical benefit was no longer met or other criteria for treatment discontinuation applied.
- Total: Total of all reporting groups
Arm/Group | Pomalidomide 0.5 mg | Placebo | China Extension: Pomalidomide 0.5 mg | Total
Number analyzed (Participants) | 168 | 84 | 15 | 267
Age, Continuous [Median (Full Range); unit: years] — Population: Results of the global study and China extension study were analyzed separately.
  years
    Global study: number analyzed (Participants) | 168 | 84 | 0 | 252
    Global study | 69.0 [40.0 to 90.0] | 69.0 [44.0 to 81.0] |  | 69.0 [40.0 to 90.0]
    China extension study: number analyzed (Participants) | 0 | 0 | 15 | 15
    China extension study |  |  | 63.0 [41.0 to 76.0] | 63.0 [41.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 28 | 6 | 75
  Male | 127 | 56 | 9 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 144 | 79 | 15 | 238
  Unknown or Not Reported | 21 | 4 | 0 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 0 | 1
  Asian | 20 | 11 | 15 | 46
  Black or African American | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islanders | 1 | 0 | 0 | 1
  White | 122 | 66 | 0 | 188
  Other | 3 | 0 | 0 | 3
  Missing | 19 | 4 | 0 | 23
Baseline RBC Transfusion Burden [Median (Inter-Quartile Range); unit: units per 28 days] — Defined as the average number of RBC-transfusion-units per 28 days over the 84 days immediately prior to randomization. Population: Data for the global study and China extension study were analyzed separately.
  units per 28 days
    Global study: number analyzed (Participants) | 168 | 84 | 0 | 252
    Global study | 2.7 [1.3 to 13.3] | 2.8 [1.3 to 10.0] |  | 2.7 [1.3 to 13.3]
    China extension study: number analyzed (Participants) | 0 | 0 | 15 | 15
    China extension study |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: -0 = Fully active, no restrictions; -1 = Restricted activity but ambulatory, able to carry out work of a light nature; -2 = Ambulatory and capable of all self-care but unable to carry out work activities; -3 = Limited self-care, confined to bed or chair more than 50% of waking hours; -4 = Completely disabled, no self-care, confined to bed or chair; -5 = Dead
  Participants
    0 (Fully active) | 53 | 22 | 5 | 80
    1 (Restricted but ambulatory) | 85 | 47 | 9 | 141
    2 (Ambulatory but unable to work) | 30 | 15 | 1 | 46
    3 (Limited self-care) | 0 | 0 | 0 | 0
    4 (Completely disabled) | 0 | 0 | 0 | 0
Disease Sub-type [Count of Participants; unit: Participants]
  Primary myelofibrosis | 127 | 65 | 10 | 202
  Post-polycythemia vera myelofibrosis | 17 | 8 | 2 | 27
  Post-essential thrombocythemia myelofibrosis | 23 | 11 | 3 | 37
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved RBC-Transfusion Independence
Description: RBC-transfusion independence was defined as the absence of RBC transfusions for any consecutive 84-day interval.
Time Frame: 168 days
Population: Global study intent to treat population (ITT) which includes all participants randomized to either of the two study drugs, regardless of whether or not any study drug was actually taken.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pomalidomide 0.5 mg: Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects or disease progression.
  Participants who were RBC-transfusion independent or experienced clinical benefit could continue to receive pomalidomide until loss of RBC-transfusion independence response or clinical benefit, or other criteria for treatment discontinuation applied.
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 168 | 84
percentage of participants | 17.3 [11.88 to 23.84] | 16.7 [9.42 to 26.38]
Statistical Analysis 1: Comparison: Pomalidomide 0.5 mg vs Placebo; Test type: Other; p = 1.000, Fisher Exact

2. Primary Outcome: China Extension: Number of Participants Achieving a Hemoglobin Increase of ≥ 15 g/L Compared to Baseline for ≥ 84 Consecutive Days
Description: A response in the China extension study was defined as an increase in hemoglobin ≥ 15 g/L above baseline value (in the absence of RBC transfusion) for ≥ 84 consecutive days.
Time Frame: From the first dose of study drug until treatment discontinuation; median treatment duration was 24.0 weeks.
Population: China extension intent-to-treat population, which includes all participants enrolled in the China extension study.
Measure: Count of Participants; unit: Participants
Groups:
- China Extension: Pomalidomide 0.5 mg: Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects, disease progression, or they received a RBC-transfusion.
Arm/Group | China Extension: Pomalidomide 0.5 mg
Number analyzed (Participants) | 15
Participants | 1

3. Secondary Outcome: Overall Survival
Description: The time from randomization to the death or to the latest date when participants are known to be alive. Overall survival was analyzed using Kaplan-Meier method; participants who were alive or lost to follow-up were censored at the latest date they were known to be alive.
Time Frame: From first dose of study drug up to end of study; median follow-up time was 19.1 months in the pomalidomide 0.5 mg arm and 17.6 months in the placebo arm.
Population: Global study intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 168 | 84
months | 24.2 [19.5 to 33.5] | 26.2 [18.0 to 32.6]
Statistical Analysis 1: Comparison: Pomalidomide 0.5 mg vs Placebo; Test type: Other; p = 0.929, Log Rank

4. Secondary Outcome: Duration of RBC-Transfusion Independence
Description: The duration of RBC-transfusion independence is the time from the date at which the first RBC-transfusion independence started to the date of another RBC-transfusion given at least 84 days after the time the transfusion independence started. The duration of the RBC-transfusion independence was analyzed using the Kaplan-Meier method. Data were censored at the end of the treatment phase for participants who had not received another RBC-transfusion after the start of transfusion independence by the end of treatment phase.
Time Frame: From first dose of study drug up to 28 days after last dose, as of the data cut-off date of 16 Jan 2013; median treatment duration was 23.6 weeks in the pomalidomide arm and 23.9 weeks in the placebo arm.
Population: Global study intent-to-treat population with an 84-day RBC-transfusion independence response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 29 | 14
months | NA [4.8 to NA] — Could not be calculated due to the low number of participants with an event | 5.8 [3.0 to NA] — Could not be calculated due to the low number of participants with an event

5. Secondary Outcome: Time to RBC-Transfusion Independence
Description: Time to response was measured from first dose of study drug to the start of the first response. The start date of the response was defined as one day after the last date of an RBC-transfusion for participants who received a RBC-transfusion after the first dose, and as the date of the first dose of study drug for participants who received no RBC-transfusions during the 84 days after the first dose of study drug.
Time Frame: 168 days
Population: Global study intent-to-treat population with an 84-day RBC-transfusion independence response
Measure: Median (Full Range); unit: weeks
Groups:
- Pomalidomide 0.5 mg: Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects or disease progression.
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 29 | 14
weeks | 6.9 [0.1 to 20.1] | 2.4 [0.1 to 15.4]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: A TEAE is an adverse event (AE) that starts on or after the first dose of study drug. The severity of each AE was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE),Version 4.0 and according to the following scale: Grade 1 = Mild (transient or mild discomfort; no limitation in activity; no medical intervention/therapy required); Grade 2 = Moderate (mild to moderate limitation in activity, some assistance may be needed; minimal medical intervention/therapy required); Grade 3 = Severe (marked limitation in activity, assistance usually required; medical intervention/therapy required, hospitalization possible); Grade 4 = Life-threatening (extreme limitation in activity, significant assistance or medical intervention/therapy required, hospitalization or hospice care probable); Grade 5 = Death Drug-related (related) AEs are those suspected by the Investigator as being related to administration of study drug
Time Frame: From the first dose of study drug until 28 days after last dose; median treatment duration was 23.7 weeks in the pomalidomide arm, 23.9 weeks in the placebo arm, and 24.0 weeks in the China extension pomalidomide arm.
Population: Participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide 0.5 mg | Placebo | China Extension: Pomalidomide 0.5 mg
Number analyzed (Participants) | 167 | 83 | 15
Participants
  Any adverse event (AE) | 164 | 81 | 12
  Adverse event suspected as related to study drug | 90 | 32 | 3
  Adverse event leading to dose interruption | 48 | 17 | 2
  Drug-related AE leading to dose interruption | 26 | 6 | 1
  AE leading to discontinuation of study drug | 53 | 14 | 0
  Related AE leading to study drug discontinuation | 21 | 8 | 0
  Grade 3/4 adverse event | 100 | 44 | 4
  Grade 3/4 AE related to study drug | 45 | 13 | 0
  Grade 3/4 AE leading to study drug discontinuation | 33 | 9 | 0
  Grade 3/4 AE leading to dose interruption | 36 | 14 | 1
  Grade 5 adverse event | 17 | 10 | 0
  Grade 5 AE related to study drug | 1 | 3 | 0
  Serious adverse event (SAE) | 76 | 29 | 0
  SAE related to study drug | 24 | 7 | 0
  SAE leading to discontinuation of study drug | 31 | 8 | 0
  SAE leading to dose interruption | 22 | 7 | 0

7. Secondary Outcome: Healthcare Resource Utilization
Time Frame: as for outcome 4
Population: Analysis of healthcare resource utilization data were not collected during the study and no analysis were performed.
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in EuroQoL-5D (EQ-5D) Health Index Score
Description: EQ-5D is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D includes 2 components: the EQ-5D health state profile (descriptive system) and the EQ-5D visual analog scale (VAS). For the health state profile participants rate their perceived health state today on 5 dimensions: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression on a Likert-type scale from 1 to 3, where 1 = "no problems," 2 = "some problems," and 3 = "extreme problems." The EQ-5D Health Utility Index (HUI) was generated from the five health state domain scores, and ranges from -0.594 (worst) and 1 (best) imaginable health state, with -0.594 representing an "unconscious" health state.
Time Frame: Baseline and Days 85 and 169
Population: Global study intent-to-treat population with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 162 | 82
score on a scale
  Day 85: number analyzed (Participants) | 112 | 56
  Day 85 | -0.0385 (0.2480) | -0.0298 (0.2129)
  Day 169: number analyzed (Participants) | 41 | 13
  Day 169 | -0.0202 (0.1666) | 0.0766 (0.1546)

9. Secondary Outcome: Change From Baseline in EuroQoL-5D (EQ-5D) Visual Analog Scale
Description: EQ-5D is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D includes 2 components: the EQ-5D health state profile (descriptive system) and the EQ-5D visual analog scale (VAS). On the VAS the participant rates his/her health state on a line from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline and Days 85 and 169
Population: Global study intent-to-treat population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 161 | 81
units on a scale
  Day 85: number analyzed (Participants) | 111 | 55
  Day 85 | 2.0 (20.78) | -1.4 (14.07)
  Day 169: number analyzed (Participants) | 41 | 13
  Day 169 | 2.9 (22.85) | 0.3 (24.25)

10. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) Total Score
Description: The FACT-An is a 47-item, cancer-specific questionnaire consisting of a core 27-item general questionnaire measuring the four general domains of QoL (physical, social/family, emotional and functional well-being), and an additional 20-item anemia questionnaire (FACT-An Anemia subscale) that measures 13 fatigue-associated items (FACT-F Fatigue subscale) and seven non-fatigue-related items. Each item is scored using a 5-point Likert rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much). FACT-An total score is calculated by adding all the FACT-An subscales together. The total score ranges from 0-188 with higher scores representing better QOL.
Time Frame: Baseline and Days 85 and 169
Population: Global study intent-to-treat population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide 0.5 mg | Placebo
Number analyzed (Participants) | 159 | 81
units on a scale
  Day 85: number analyzed (Participants) | 109 | 56
  Day 85 | -2.1 (20.32) | 4.3 (18.73)
  Day 169: number analyzed (Participants) | 41 | 13
  Day 169 | 6.2 (20.49) | 11.9 (18.60)

ADVERSE EVENTS:
Time Frame: All-cause mortality data are reported from first dose of study drug up to end of study; maximum follow-up time was 85 months. Adverse events are reported from the first dose of study drug until 28 days after last dose; median treatment duration was 23.7 weeks in the pomalidomide arm, 23.9 weeks in the placebo arm, and 24.0 weeks in the China extension pomalidomide arm.
Description: The safety population includes all participants who received at least one dose of study drug; one participant randomized to pomalidomide and one participant randomized to placebo in the global study did not receive treatment and are excluded from the safety population.
Groups:
- Global Study: Pomalidomide 0.5 mg: Participants received pomalidomide 0.5 mg/day by mouth for at least 168 days unless there were unacceptable side effects or disease progression. Participants who experienced clinical benefit (defined as a reduction from Baseline of ≥ 50% in RBC-transfusion frequency during the prior 84-day interval) could continue to receive pomalidomide until the definition of clinical benefit was no longer met or other criteria for treatment discontinuation applied.
- Global Study: Placebo: Participants received placebo taken by mouth once daily for at least 168 days unless there were unacceptable side effects or disease progression. Participants who experienced clinical benefit could continue to receive placebo until the definition of clinical benefit was no longer met or other criteria for treatment discontinuation applied.
Arm/Group | Global Study: Pomalidomide 0.5 mg | Global Study: Placebo | China Extension: Pomalidomide 0.5 mg
All-Cause Mortality (participants affected / at risk) | 115/167 | 54/83 | 8/15
Serious Adverse Events (participants affected / at risk) | 76/167 | 29/83 | 0/15
Other Adverse Events (participants affected / at risk) | 155/167 | 76/83 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Global Study: Pomalidomide 0.5 mg (N=167) | Global Study: Placebo (N=83) | China Extension: Pomalidomide 0.5 mg (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 10 | 3 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 1 | 0
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
SPLENIC EMBOLISM (Blood and lymphatic system disorders) | 1 | 0 | 0
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 1 | 0
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 2 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 2 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 5 | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 0 | 0
CONDUCTION DISORDER (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
ASTHENIA (General disorders) | 2 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 2 | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 4 | 0 | 0
PYREXIA (General disorders) | 5 | 3 | 0
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1 | 0
SUDDEN DEATH (General disorders) | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 0 | 0
BACTEROIDES BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
GASTROINTESTINAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 3 | 1 | 0
LYMPHADENITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
NECROTISING FASCIITIS (Infections and infestations) | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 6 | 4 | 0
SEPSIS (Infections and infestations) | 1 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 0
SIALOADENITIS (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 1 | 0
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TRANSFUSION-RELATED CIRCULATORY OVERLOAD (Injury, poisoning and procedural complications) | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0
PLATELET COUNT INCREASED (Investigations) | 0 | 1 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
HISTIOCYTOSIS HAEMATOPHAGIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 3 | 0
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 1 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 | 0 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
PHLEBITIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Global Study: Pomalidomide 0.5 mg (N=167) | Global Study: Placebo (N=83) | China Extension: Pomalidomide 0.5 mg (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 12 | 5 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 25 | 4 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 21 | 12 | 1
ARRHYTHMIA (Cardiac disorders) | 2 | 1 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 11 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 22 | 11 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 | 3 | 0
CONSTIPATION (Gastrointestinal disorders) | 24 | 9 | 0
DIARRHOEA (Gastrointestinal disorders) | 35 | 17 | 2
NAUSEA (Gastrointestinal disorders) | 21 | 16 | 0
VOMITING (Gastrointestinal disorders) | 12 | 7 | 0
ASTHENIA (General disorders) | 23 | 8 | 0
CHEST PAIN (General disorders) | 2 | 0 | 1
FATIGUE (General disorders) | 35 | 17 | 3
OEDEMA (General disorders) | 1 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 53 | 14 | 1
PYREXIA (General disorders) | 30 | 9 | 2
HEPATIC CYST (Hepatobiliary disorders) | 1 | 0 | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 9 | 4 | 2
NASOPHARYNGITIS (Infections and infestations) | 13 | 0 | 0
PNEUMONIA (Infections and infestations) | 10 | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 5 | 1
URINARY TRACT INFECTION (Infections and infestations) | 12 | 2 | 0
FALL (Injury, poisoning and procedural complications) | 7 | 5 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 1
WEIGHT DECREASED (Investigations) | 11 | 3 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 | 0 | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 20 | 7 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 2 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 7 | 5 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 8 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9 | 5 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 6 | 0
DIZZINESS (Nervous system disorders) | 17 | 12 | 0
SOMNOLENCE (Nervous system disorders) | 5 | 5 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 24 | 9 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 28 | 8 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 10 | 3 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 12 | 5 | 0
RASH (Skin and subcutaneous tissue disorders) | 11 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then Investigator can publish if the manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides a publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.